CLINICAL TRIAL: NCT04674631
Title: The Effect of Neuropathic Pain on Quality of Life, Depression and Sleep in Patients With Combat-related Extremity Injury
Brief Title: The Effect of Neuropathic Pain in Patients With Combat-related Extremity Injury
Status: Completed | Type: Observational
Sponsor: Gaziler Physical Medicine and Rehabilitation Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Yasin Demir, Physical Medicine and Rehabilitation Associate Professor, Gaziler Physical Medicine and Rehabilitation Education and Research Hospital
Other Study IDs: 8
Record Dates: First submitted 2020-12-14; First posted 2020-12-19 (Actual); Last update posted 2021-12-02 (Actual); Status verified 2021-11

CONDITIONS: Neuropathic Pain
MeSH Terms: conditions — Neuralgia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case group 1: 52 patients with score of 12 or more on Leeds assessment of neuropathic symptoms and signs (LANSS) questionnaire will be included in the neuropathic pain group.
  Interventions: Other: The effect of neuropathic pain on quality of life, depression and sleep quality
- Case group 2: 46 patients with scores less than 12 on LANSS will be included in the group without neuropathic pain.
  Interventions: Other: The effect of neuropathic pain on quality of life, depression and sleep quality

INTERVENTIONS:
Other: The effect of neuropathic pain on quality of life, depression and sleep quality — The effect of neuropathic pain on quality of life, depression and sleep quality

SUMMARY:
It has been suggested that veterans with chronic pain might be at increased risk for the development of depression, anxiety and post-traumatic stress disorder. To date, most of the published studies have focused on chronic pain as a whole, and there are limited studies examining association of neuropathic pain with psychological comorbidity and quality of life.Combat related extremity injury significantly influences the patients' quality of life and psychological state. In this context, the purpose of this study is to illustrate to what extent neuropathic pain influences the quality of life, depression level and sleep quality of patients with combat-related extremity injury.

DETAILED DESCRIPTION:
A total of 120 patients with combat-related extremity injury and 60 age and BMI-matched healthy controls will be participated in this cross-sectional study. The presence of neuropathic pain will be evaluated using Leeds assessment of neuropathic symptoms and signs (LANSS) questionnaire. The impact of pain on health-related quality of life will be assessed using the 36-Item Short Form Survey (SF-36). Beck Depression Scale (BDS) will be used to evaluate depression status of the patients. Quality of sleep will be assessed using the Pittsburgh Sleep Quality Index (PSQI).

ELIGIBILITY:
Inclusion Criteria:

* Patients between the ages of 18-65 years who had previous history of combat-related extremity injury

Exclusion Criteria:

* Previous history of the cervical or lumbosacral radiculopathy, any known rheumatic disease or neurologic or endocrine disorders, excessive alcohol consumption and vitamin B12 deficiency

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A total of 98 patients with combat-related extremity injury
Sampling Method: Probability Sample
Enrollment: 98 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2021-11-01 (Actual)

PRIMARY OUTCOMES:
Short Form Survey (SF-36) | through study completion, an average of one and a half months
  The impact of pain on health-related quality of life will be assessed using the 36-Item Short Form Survey (SF-36). The validity and reliability of the Turkish version of SF-36 has been illustrated. SF-36 is a common questionnaire for the evaluation of quality of life, and it includes a total of 36 items in eight separate scales (physical functioning, general health, physical role, bodily pain, vitality, social functioning, mental health and emotional role). Each subscale is scored between 0 and 100, and high scores indicate better quality of life
Beck Depression Scale (BDS) | through study completion, an average of one and a half months
  Beck Depression Scale (BDS) will be used to evaluate depression status of the patients. Beck Depression Scale, which is a 21-item self report rating inventory, measures characteristic symptoms and attitudes of depression. The scale is scored between 0 and 63. The cut-off point considered is 17. Higher scores reflect more severe depression.
Pittsburgh Sleep Quality Index (PSQI) | through study completion, an average of one and a half months
  Quality of sleep will be assessed using the Pittsburgh Sleep Quality Index (PSQI), which assesses the individual's self-reported quality of sleep during the last month [9]. This 19-item index evaluates seven components of quality of sleep: subjective quality of sleep, sleep duration, sleep latency, sleep disturbances, sleep efficiency, drug use for sleep, and daytime dysfunction. A total PSQI score (range, 0-21) is the total of particular scores from the seven components. A score of ≥6 is considered to indicate poor quality of sleep. The Turkish validation of PSQI was performed.

CONTACTS AND LOCATIONS:
Overall Officials: Merve Orucu Atar, MD, Principal Investigator — Gaziler PMR, Training and Research Hospital, Department of PMR
Locations (1):
- Merve Orucu Atar, Ankara, Cankaya, Turkey (Türkiye)